CLINICAL TRIAL: NCT00485901
Title: A Double-Blind Randomized Comparison of the Efficacy and Safety of Intramuscular Olanzapine and Intramuscular Haloperidol in Acutely Agitated Patients With Schizophrenia
Brief Title: Comparison of Intramuscular Olanzapine and Intramuscular Haloperidol in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6409; F1D-TW-S025
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — olanzapine-fluoxetine combination; Haloperidol

INTERVENTIONS:
Drug: Olanzapine Hydrochloride
Drug: Haloperidol

SUMMARY:
The purpose of this study is to compare intramuscular Olanzapine and intramuscular Haloperidol in changing of agitation in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, between the ages of 18 and 65
* Patients must have diagnosis of schizophrenia that meets disease diagnostic criteria as defined in DSM-IV
* Patients must be considered, by the investigator, to be clinically agitated and appropriate candidates for treatment with IM medication. Investigator must believe that it is safe to administer IM olanzapine and IM comparator to the patients with respect to the safety profile of these drugs (including the anticholinergic properties of Olanzapine IM or the comparator agent)
* Subjects' illness must not, in the opinion of the investigator, be caused by substance abuse
* Patient must be hospitalized during the study

Exclusion Criteria:

* Previous participation (treatment with study drug) in a Lilly sponsored intra-muscular olanzapine clinical trial
* Serious, unstable illnesses such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months
* Have a known diagnosis of dementia of any type, as defined in the DSM-IV or DSM-IV-TR
* Documented history of allergic reaction to study medication(s)
* Treatment with an injectable depot neuroleptic within 1 injection interval prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of IM olanzapine compared with IM haloperidol in changing of agitation from baseline to 2 hours post-first IM injection

SECONDARY OUTCOMES:
Assess treatment-emergent adverse events, change in vital signs and extrapyramidal symptoms of IM olanzapine versus IM haloperidol during the study
Assess the efficacy of IM olanzapine compared with IM haloperidol from baseline to 15 min, 30 min, 60 min and 120 minutes post-first IM injection
Compare the response rates and time to response during the 2 hours post-first IM injection.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei, Taiwan

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com